CLINICAL TRIAL: NCT06846541
Title: An Extension Study in Patients With Moderate to Severe Plaque Psoriasis to Evaluate the Long-term Safety, Efficacy, and Durability of Response to ESK-001
Brief Title: Long-term Safety and Efficacy of ESK-001 in Moderate to Severe Plaque Psoriasis
Acronym: ONWARD3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESK-001-018
Record Dates: First submitted 2025-01-27; First posted 2025-02-26 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Plaque Psoriasis; Psoriasis (PsO); Psoriasis; Moderate Psoriasis; Severe Psoriasis
Keywords: Psoriasis; PASI; Safety; ESK-001
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Open-Label ESK-001 (Experimental): Open-Label ESK-001 administered as an oral tablet
  Interventions: Drug: Open-Label ESK-001
- Blinded ESK-001 (Experimental): Blinded ESK-001 administered as an oral tablet
  Interventions: Drug: Blinded ESK-001
- Placebo (Placebo Comparator): Matching placebo administered as an oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Open-Label ESK-001 — Open-Label ESK-001
  Arms: Open-Label ESK-001
Drug: Blinded ESK-001 — Blinded ESK-001 during Randomized Treatment Withdrawal Period
  Arms: Blinded ESK-001
Drug: Placebo — Placebo during Randomized Treatment Withdrawal Period
  Arms: Placebo

SUMMARY:
The objective of the ESK-001-018 long term extension is to evaluate the safety and efficacy of ESK-001 over time. The scientific questions it aims to answer are:

* How safe is taking ESK-001 long-term in people with moderate to severe plaque psoriasis?
* Does taking ESK-001 long-term reduce the severity of people's plaque psoriasis?

Patients will enter the long-term extension study following completion of one of the parent studies (ESK-001-016 or ESK-001-017) and will receive open-label ESK-001 twice daily for 24 weeks. After 24 weeks, the first 200 patients meeting at least PASI-75 clinical response will be randomly assigned to receive ESK-001 or placebo. At any point during this time, the patients losing the initial clinical response may return to the open-label ESK-001 treatment. Patients who complete Week 48 will return to open-label ESK-001 treatment and they will receive ESK-001 until the end of the study or discontinuation. All the remaining patients not meeting the entry criteria for the randomized withdrawal phase will continue to receive open-label ESK-001 for the remainder of the study.

Patients taking part in the study must be men or women aged at least 18 years old and have completed a previous (parent) study of ESK-001 in moderate to severe plaque psoriasis.

Patients must consent and agree to:

* ensure drug daily compliance until end of study or discontinuation.
* visit the clinic for checkups and assessments.
* provide blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age ≥18 years
2. Completed either of the two previous (parent) studies of ESK-001 (ESK-001-016 or ESK-001-017)
3. ESK-001 safety and tolerability were acceptable in the parent study
4. Women of childbearing potential (WOCBP) and males who are sexually active with WOCBP must agree to adhere to highly effective methods of contraception for the entirety of the study

Exclusion Criteria:

1. Pregnant, lactating, or planning to get pregnant during the study period
2. Any acute or chronic illness/condition or evidence of an unstable clinical condition that in the Investigator's judgment will substantially increase the risk to the patient if they continue to receive ESK-001 treatment in this extension study
3. Deemed by the Investigator to be inappropriate for the study or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1680 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To assess the long-term safety and tolerability of ESK-001 throughout the duration of the study | Approximately 4 years
  Incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
To assess the long-term efficacy of ESK-001 using the Psoriasis Area and Severity Index (PASI-75) | 24, 48, 72, and 96 weeks
  Proportion of patients achieving ≥75% reduction in PASI
To assess the long-term efficacy of ESK-001 using the Psoriasis Area and Severity Index (PASI-90) | 24, 48, 72, and 96 weeks
  Proportion of patients achieving ≥90% reduction in PASI
To assess the long-term efficacy of ESK-001 using the Psoriasis Area and Severity Index (PASI-100) | 24, 48, 72, and 96 weeks
  Proportion of patients achieving 100% reduction in PASI
To assess the long-term efficacy of ESK-001 using the Static Physician's Global Assessment (sPGA 0/1) | 24, 48, 72, and 96 weeks
  Proportion of patients achieving a score of 0 or 1 on sPGA
To assess the long-term efficacy of ESK-001 based on change in Psoriasis Area and Severity Index (PASI) | 24, 48, 72, and 96 weeks
  Change in Psoriasis Area and Severity Index (PASI) from baseline assessments
To assess the long-term efficacy of ESK-001 based on change in Affected Body Surface Area (%BSA) | 24, 48, 72, and 96 weeks
  Change in affected body surface area (%BSA) from baseline assessments
To characterize the loss of PASI-75 response following withdrawal of ESK-001 treatment (only for patients randomized to the treatment withdrawal phase) | Week 48
  Median time to loss of PASI-75 response
To characterize the loss of PASI-90 response following withdrawal of ESK-001 treatment (only for patients randomized to the treatment withdrawal phase) | Week 48
  Median time to loss of PASI-90 response
To characterize the loss of sPGA-0/1 response following withdrawal of ESK-001 treatment (only for patients randomized to the treatment withdrawal phase) | Week 48
  Median time to loss of sPGA-0/1 response
To assess the change in quality of life (QoL) using Dermatology Life Quality Index after long-term ESK-001 administration | Week 24, Week 48, and Week 72
  Proportion of patients achieving a DLQI-0/1 score of 0 (no effect) or 1 (minimal effect)

CONTACTS AND LOCATIONS:
Locations (268):
- United States (92):
  - Total Dermatology, Birmingham, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Alliance Dermatology, Pheonix, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Northwest AR Clinical Trials Center PLLC, Rogers, Arkansas
  - Zenith Research Inc., Beverly Hills, California
  - Exalt Clinical Research Inc, Chula Vista, California
  - California Dermatology and Clinical Research Institute, Encinitas, California
  - Raoof MD, Encino, California
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Marvel Clinical Research LLC, Huntington Beach, California
  - Long Beach Research Institute, Long Beach, California
  - Olive View UCLA Education and Research Institute, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Wallace Medical Group Inc, Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - Pasadena Clinical Trials, Pasadena, California
  - Empire Clinical Research Pomona, Pomona, California
  - Integrative Skin Science and Research, Sacramento, California
  - Therapeutics Clinical Research, San Diego, California
  - Southern California Clinical Research, Santa Ana, California
  - Clinical Science Institute Dermatology Institute, Santa Monica, California
  - Unison Clinical Trials, Sherman Oaks, California
  - California Dermatology Institute Thousand Oaks, Thousand Oaks, California
  - Sunwise Clinical Research LLC, Walnut Creek, California
  - Clearlyderm Dermatology West Boca Raton, Boca Raton, Florida
  - Driven Clinical Research, Coral Gables, Florida
  - FXM Clinical Research Ft. Lauderdale LLC, Fort Lauderdale, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Glick Skin Institute, Margate, Florida
  - AppleMed Research Group, Miami, Florida
  - FAX Pharma Clinical Research Inc, Miami, Florida
  - FXM Clinical Research Miami LLC, Miami, Florida
  - Las Mercedes Medical Research, Miami, Florida
  - Procare Research Center, Miami Gardens, Florida
  - San Marcus Research Clinic Inc - Miami, Miami Lakes, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - FXM Clinical Research Miramar LLC, Miramar, Florida
  - Oceanic Research Group, North Miami Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Lenus Research and Medical Group LLC, Sweetwater, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - ForCare Medical Center, Tampa, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - NorthShore Medical Group Dermatology Skokie, Skokie, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - DS Research of Southern Indiana, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, Columbus, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Equity Medical, Bowling Green, Kentucky
  - DS Research of Kentucky, Louisville, Kentucky
  - Velocity Clinical Research, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MetroBoston Clinical Partners, Brighton, Massachusetts
  - Michigan Center for Research Company, Clarkston, Michigan
  - Henry Ford Medical Center Farmington, Detroit, Michigan
  - Revival Research Institute, Troy, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Associated Skin Care Specialists Minnesota Clinical Study Center, New Brighton, Minnesota
  - Cleaver Dermatology, Kirksville, Missouri
  - Schlessinger MD, Omaha, Nebraska
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - NYC Health and Hospitals Elmhurst, Elmhurst, New York
  - Pioneer Clinical Research NY, New York, New York
  - Cameron Dermatology, New York, New York
  - OptiSkin, New York, New York
  - DermResearchCenter of New York, Stony Brook, New York
  - Asheville Clinical Trials, Asheville, North Carolina
  - WDC Cosmetic and Research, Wilmington, North Carolina
  - Optima Research Boardman, Boardman, Ohio
  - The Ohio State University Wexner Medical Center OSUWMC OSU Dermatology East Columbus, Gahanna, Ohio
  - Dermatologists of Southwestern Ohio LLC, Mason, Ohio
  - Unity Clinical Research UCR, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Medford, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Clinical Partners LLC, Johnston, Rhode Island
  - Studies in Dermatology LLC, Cypress, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Reveal Research Institute, Frisco, Texas
  - Center for Clinical Studies Texas Medical Center, Houston, Texas
  - Austin Institute for Clinical Research, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Progressive Clinical Research San Antonio, San Antonio, Texas
  - Center for Clinical Studies (CCS) - Webster/Clear Lake Location, Webster, Texas
  - University of Utah Health Care Midvalley Health Center, Murray, Utah
  - Jordan Valley Dermatology, South Jordan, Utah
  - Frontier Dermatology, Mill Creek, Washington
- Australia (4):
  - Premier Specialist, Kogarah, New South Wales
  - North Eastern Health Specialists, Campbelltown, South Australia
  - Skin Health Institute, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment Dr Tota Venkova, Gabrovo
  - Medikal Center Kordis, Pleven
  - Skin and Venereal Diseases Center EOOD, Sofia
  - DCC Aleksandrovka, Sofia
  - University Multiprofile Hospital for Active Treatment Alexandrovska, Sofia
- Canada (29):
  - Rejuvenation Medical Group Edmonton Downtown, Edmonton, Alberta
  - Alberta DermaSurgery, Edmonton, Alberta
  - VIDA Dermatology/VIDA Clinical Research, Edmonton, Alberta
  - CaRe Clinic Red Deer, Red Deer, Alberta
  - Enverus Medical, Surrey, British Columbia
  - CCA Medical Research Corp, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - SKiN Health, Coburg, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Dermatrials Research Inc, Hamilton, Ontario
  - Centricity Research London, London, Ontario
  - Derm Effects, London, Ontario
  - Lynderm Research, Markham, Ontario
  - DermEdge Research Inc, Mississauga, Ontario
  - Clear Skin Dermatology, Newmarket, Ontario
  - North Bay Dermatolgy Centre, North Bay, Ontario
  - Canadian Dermatology Centre, North York, Ontario
  - Rejuvenation Dermatology - Oakville, Oakville, Ontario
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - North York Research Inc, Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Dermatology on Bloor, Toronto, Ontario
  - Alliance Clinical Trials Inc, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Innovaderm, Montreal, Quebec
  - Centre of Research in Dermatology Quebec CRDQ, Québec, Quebec
  - Dermatologie Sima Inc, Verdun, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- Czechia (15):
  - Dermamedica, Náchod, Královéhradecký kraj
  - Vesalion s.r.o, Ostrava, Moravian Silesian
  - Sanatorium Profesora Arenbergera, Prague, Prague
  - Clintrial sro, Prague, Prague
  - Pratia Brno, Brno
  - Lékárna Pod Kaňkem, Kutná Hora
  - Nemocnice Novy Jicin, Nový Jičín
  - Dermskin sro, Olomouc
  - CCR Ostrava, Ostrava
  - Pratia Pardubice as, Pardubice
  - Fakultni nemocnice Plzen Dermatovenerologicka klinika, Pilsen
  - Fakultni Nemocnice Kralovske Vinohrady FNKV Dermatovenerologicka Klinika, Prague
  - Pratia Prague, Prague
  - Praglandia, Prague
  - Dermatologicka ambulance Svitavy, Svitavy
- Estonia (4):
  - Innomedica, Tallinn, Harju
  - Tartu University Hospital, Tartu, Tartu
  - Center for Clinical and Basic Research AS, Tallinn
  - Kliiniliste Uuringute Keskus OU, Tartu
- France (2):
  - Centre Azur Nice, Nice, Alpes Maritimes
  - CHU de Rouen, Rouen, Essais Cliniques
- Germany (23):
  - Hautarztpraxis Dr Mihaescu, Augsburg, Augsburg
  - Eberhard Karls Universitaet Tuebingen Universitaets Hautklinik Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitatsklinikum Erlangen, Erlangen, Bavaria
  - Hautarztpraxis Mahlow, Mahlow, Brandenburg
  - Rosenpark Research, Darmstadt, Hesse
  - Universitatsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Hautarztpraxis an der Hase, Bramsche, Lower Saxony
  - Klinikum Oldenburg, Oldenburg, Lower Saxony
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Klinikum Bielefeld, Bielefeld, North Rhine-Westphalia
  - Hautarztpraxis Dr Niesmann and Dr Othlinghaus, Bochum, North Rhine-Westphalia
  - Intramedis CSS, Remscheid, North Rhine-Westphalia
  - Dermatologische Praxis Dres Quist, Mainz, Rhinelkand-Palatinate
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - Praxis fur Dermatologie und Venerologie, Dresden, Saxony
  - Haut Ambulatorium Magdeburg, Magdeburg, Saxony-Anhalt
  - Universitatsklinikum Schleswig Holstein, Kiel, Schleswig-Holstein
  - MVZ DermaKiel GmbH, Kiel, Schleswig-Holstein
  - Universitatsklinikum Schleswig Holstein, Lübeck, Schleswig-Holstein
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Universitaetsklinikum Muenster, Münster
  - KliFOs Klinische Forschung Osnabruck, Osnabrück
- Hungary (8):
  - Bacs Kiskun County Teaching Hospital, Kecskemét, Bács-Kiskun county
  - Bőrgyógyászati Klinika, Debreceni Egyetem Orvos - és Egészségtudományi Centrum, Debrecen, Hajdú-Bihar
  - Allergo-Derm Bakos Kft, Szolnok, JN
  - DermaMed Research Kf, Békés, Oroshaza
  - UNO Medical Trials Kft., Budapest
  - Orvostudomanyi Kutato es Fejleszto Kft, Debrecen
  - DERMA B Kft, Debrecen
  - Medmare Bt, Veszprém
- Japan (20):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Tokyo Medical University Ibaraki Medical Center, Ibaraki, Inashiki-gun
  - Saruwatari Dermatology Clinic, Kagoshima, Kagoshima-Shi
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa-shi
  - Kanto Rosai Hospital, Kanagawa, Kawasaki-shi
  - Mie University Hospital, Tsu, Mie-ken
  - Okayama University Hospital, Okayama, Okayama-shi
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka-shi
  - Nippon Life Hospital, Osaka, Osaka-Shi
  - Hokkaido University Hospital, Hokkaido, Sapporo-shi
  - Kindai University Hospital, Osaka, Sayama-Shi
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-Ku
  - Nihon University Itabashi Hospital, tabashi City, Tokyo
  - Medical Corporation Jitai kai Tachikawa Dermatology Clinic, Tachikawa, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
- Latvia (7):
  - Semigallia Ltd, Kuldīga, Kuldigas
  - Riga 1st Hospital, Riga, Rīga
  - SIA Veseliba un estetika, Riga, Rīga
  - Smite Aija medical practice in dermatology venereology, Talsi, Talsi
  - Med Art clinic, Riga
  - Veselibas Centrs 4, Riga
  - Veselibas Centrs 4 Filiale Dermatologijas Klinika, Riga
- Poland (39):
  - Specderm, Podlaski, Bialystok
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Synexus Centrum Medyczne Osteomed Wroclaw, Wroclaw, Lower Silesian Voivodeship
  - WroMedica, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne dr Rajzer spolka zoo, Krakow, Malopolska
  - Diamond Clinic, Krakow, Malopolska
  - RCMed Oddział Sochaczew, Sochaczew, Masovian Voivodeship
  - FutureMeds Warszawa Centrum, Warsaw, Masovian Voivodeship
  - Clinical Best Solutions, Warsaw, Masovian Voivodeship
  - MICS Medical Center Warsaw, Warsaw, Masovian Voivodeship
  - High Med Przychodnia Specjalistyczna, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park, Warsaw, Masovian Voivodeship
  - RoyalDerm, Warsaw, Mazowiecke
  - ClinicMed Daniluk Nowak SpK, Bialystok, Podlaskie Voivodeship
  - AES Gdansk, Gdansk, Pomeranian Voivodeship
  - Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - Derm Art Institute, Gdynia, Pomeranian Voivodeship
  - Synexus Sp zo o Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - Centrum Badan Klinicznych PI House, Gdansk, Poneranian
  - Pratia Katowice, Katowice, Silesian Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Research Solutions, Katowice, Silesian Voivodeship
  - Laser Clinic, Szczecin, West Pomeranian Voivodeship
  - Care Clinic Katowice, Katowice
  - Centrum Medyczne All Med Badania Kliniczne, Krakow
  - Pratia MCM Krakow, Krakow
  - Krakowskie Centrum Medyczne, Krakow
  - Luxderm, Lublin
  - Zanamed Medical Clinic Sp z o o, Lublin
  - Klinika Dermatologii Uniwersytecki Szpital Kliniczny im F Chopina, Rzeszów
  - Rheuma Medicus, Warsaw
  - MTZ Clinical Research Sp z o o, Warsaw
  - Centrum Medyczne Synexus Warszawa, Warsaw
  - Klinika Ambroziak Dermatologia Kliniczna, Warsaw
  - dermMedica, Wroclaw
  - Dermoklinika, Lodz, Łódź Voivodeship
  - FutureMeds Lodz, Lodz, Łódź Voivodeship
  - Velocity Clinical Research Skierniewice, Skierniewice, Łódź Voivodeship
- Portugal (3):
  - Hospital da Senhora da Oliveira, Guimarães, Braga District
  - Hospital CUF Descobertas, Lisbon, Lisbon District
  - Unidade Local de Saude Santo Antonio Hospital de Santo Antonio, Porto
- Puerto Rico (4):
  - Centro Reumatologico de Cagus, Caguas, Puerto Rico
  - Ponce Medical School Foundation Inc, Ponce, Puerto Rico
  - Clinical Research Puerto Rico, San Juan, Puerto Rico
  - GCM Medical Group PSC Hato Rey Site, San Juan
- South Korea (6):
  - Pusan National University Hospital, Seogu, Busan
  - Chosun Universtiy Hospital, Gwangju, Dong-gu
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
- Spain (7):
  - University General Hospital Dr Balmis, Alicante, Alicante
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, A Coruña, Santiago de Compostela
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital de Manises, Manises

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor Alumis Inc. is a clinical-stage biopharmaceutical company that has not yet adopted an Individual Participant Data (IPD) sharing plan.